CLINICAL TRIAL: NCT00369902
Title: Pilot Study on the Effect of Acupuncture Treatment on Pain Perception and on the Ability to Cope With Pain
Brief Title: The Effect of Acupuncture Treatment on the Perception of Pain and Coping With Pain
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: SHEBA-05-3817-OG-CTIL
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Pain
Keywords: pain; acupuncture
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: acupuncture

SUMMARY:
The Purpose of this study is to evaluate whether cognitive and emotional components take part in the positive acupuncture effect on pain.

DETAILED DESCRIPTION:
The effect of acupuncture on pain intensity has been already investigated and confirmed. Recent publication (Pariente J., et a., 2005) indicated that acupuncture may affect midbrain areas, that are associated with cognitive control of pain.

The Pain Self Regulation Model (Levental, 1980)distinguishes between emotional response pain representations and cognitive pain representations. According to this model, emotional and cognitive pain representations leads to a new (cognitive or emotional) evaluation of the pain, that affects its perception and the ability to cope with it (Levental at al., 2001).

This study will try to assess the hypothesis that acupuncture treatment is involved in this process.

The study is designed as pilot study, limited to 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from pain,who are reffered for acupuncture treatment,and consented to participate in this study

Exclusion Criteria:

* children under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 41 consequtive patients with chronic musculosckeletal pain
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Gamus, M.D., Ph.D., Principal Investigator — Sheba Hospital, Tel Hashomer, ISRAEL
Locations (1):
- Sheba Hospital,, Ramat Gan, Israel